CLINICAL TRIAL: NCT07008235
Title: Effect of Amitriptyline and Trifluoperazine on Patients With Functional Dyspepsia
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Md. Moktadirul Hoque Shuvo (Other)
Responsible Party: Sponsor-Investigator, Md. Moktadirul Hoque Shuvo, Principal Investigator, Dhaka Medical College
Organization: Dhaka Medical College (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB-DMC/2025/38
Record Dates: First submitted 2025-05-24; First posted 2025-06-06 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Functional Dyspepsia
Keywords: Functional Dyspepsia; Amitriptyline; Trifluoperazine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Amitriptyline (Active Comparator): Tab. Amitriptyline 10 milligrams at night along with first line treatment for 8 weeks after randomization. After that, the amitriptyline will be discontinued, and patients will be kept on first line treatment only for additional 4 weeks.
  Interventions: Drug: Tablet Amitriptyline 10 milligrams
- Trifluoperazine (Active Comparator): Tab. Trifluoperazine 1 milligrams twice daily along with first line treatment for 8 weeks after randomization. After that, the trifluoperazine will be discontinued, and patients will be kept on first line treatment only for additional 4 weeks.
  Interventions: Drug: Tablet Trifluoperazine 1 milligrams twice daily
- Control Group (No Intervention): First line treatment only for 12 weeks

INTERVENTIONS:
Drug: Tablet Amitriptyline 10 milligrams — Tablet Amitriptyline 10 milligrams at night will be given to patients along with standard first line treatment of functional dyspepsia for 8 weeks after randomization. After that, the amitriptyline will be discontinued, and patients will be kept on first line treatment only for additional 4 weeks.
  Arms: Amitriptyline
Drug: Tablet Trifluoperazine 1 milligrams twice daily — Tablet Trifluoperazine 1 milligrams twice daily will be given to patients along with standard first line treatment of functional dyspepsia for 8 weeks after randomization. After that, the trifluoperazine will be discontinued, and patients will be kept on first line treatment only for additional 4 weeks.
  Arms: Trifluoperazine

SUMMARY:
The goal of this clinical trial is to assess and compare the effect of amitriptyline and trifluoperazine in improving dyspeptic symptoms in patients with functional dyspepsia. It will also assess about the safety of drugs amitriptyline and trifluoperazine by recording the patient reported adverse events. The main questions it aims to answer are:

Does drug amitriptyline and trifluoperazine has any effect on patients with functional dyspepsia? What medical problems do participants have when taking drug amitriptyline and trifluoperazine? Researcher will compare drug amitriptyline and trifluoperazine to a control group taking standard first line treatment only.

Participants will:

Take drug amitriptyline 10 milligrams at night or trifluoperazine 1 milligrams twice daily every day for 8 weeks along with standard first line treatment. A third group will be taken as control arm who will be kept on standard first line treatment only for 8 weeks. After that all three groups will be kept only on standard first line treatment for an additional 4 weeks. They will visit the hospital 4 weekly, and their symptoms will be assessed by a 5-point Likert Scale at baseline, week 4, 8, and 12. Additionally, patient reported adverse events will be documented.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or more
* Patients with symptoms of dyspepsia for duration consisted with ROME IV criteria
* Patients who are willing to sign informed written consent

Exclusion Criteria:

* Structural lesion in Upper GI endoscopy and/or positive CLO test
* Patients scoring 1 or 2 on the 5-point Likert scale for all four dyspepsia symptoms
* History of malignancy, significant liver and biliary tract disease, hypertension, diabetes mellitus, chronic kidney disease, thyroid disorder, major psychiatric disorders
* Previous history of gastrointestinal surgery
* Patients those have to take any drug for other medical condition that may cause dyspepsia
* Any patient with ongoing treatment with antidepressants or antipsychotics
* Any history of hypersensitivity, adverse effect, or ineffectiveness with amitriptyline or trifluoperazine
* Patients for whom Amitriptyline and Trifluoperazine are contraindicated
* Elderly patients> 60 years
* Pregnancy and breastfeeding

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Change in dyspeptic symptom | At baseline and then at week 4 and 8 after randomization
  The change of four dyspeptic symptoms (Postprandial fullness, Early Satiety, Epigastric pain, Epigastric burning) will be assessed by a 5-point Likert Scale. The four main symptoms of dyspepsia, each will be graded as 1 (No problem), 2 (Mild problem, can be ignored when not thinking about it), 3 (Moderate problem, cannot be ignored but does not influence daily activities), 4 (Severe Problem, influences concentration on daily activities), 5 (Very severe problem, markedly influences daily activities or requires rest or both). The total minimum value is 4 and maximum value is 20. Higher score means worse outcome.

SECONDARY OUTCOMES:
See the effect of trifluoperazine compared to first line treatment only | At baseline and then at week 4 and 8 after randomization
  Effect of trifluoperazine on four dyspeptic symptoms (Postprandial fullness, Early Satiety, Epigastric pain, Epigastric burning) will be assessed and compared to first line treatment only by a 5-point Likert Scale. The four main symptoms of dyspepsia, each will be graded as 1 (No problem), 2 (Mild problem, can be ignored when not thinking about it), 3 (Moderate problem, cannot be ignored but does not influence daily activities), 4 (Severe Problem, influences concentration on daily activities), 5 (Very severe problem, markedly influences daily activities or requires rest or both). The total minimum value is 4 and maximum value is 20. Higher score means worse outcome.
See the effect of amitriptyline compared to first line treatment only | At baseline and then at week 4 and 8 after randomization
  Effect of amitriptyline on four dyspeptic symptoms (Postprandial fullness, Early Satiety, Epigastric pain, Epigastric burning) will be assessed and compared to first line treatment only by a 5-point Likert Scale. The four main symptoms of dyspepsia, each will be graded as 1 (No problem), 2 (Mild problem, can be ignored when not thinking about it), 3 (Moderate problem, cannot be ignored but does not influence daily activities), 4 (Severe Problem, influences concentration on daily activities), 5 (Very severe problem, markedly influences daily activities or requires rest or both). The total minimum value is 4 and maximum value is 20. Higher score means worse outcome.
Compare the effects of amitriptyline and trifluoperazine | At baseline and then at week 4 and 8 after randomization
  Effect of amitriptyline and trifluoperazine on four dyspeptic symptoms (Postprandial fullness, Early Satiety, Epigastric pain, Epigastric burning) will be assessed and compared by a 5-point Likert Scale. The four main symptoms of dyspepsia, each will be graded as 1 (No problem), 2 (Mild problem, can be ignored when not thinking about it), 3 (Moderate problem, cannot be ignored but does not influence daily activities), 4 (Severe Problem, influences concentration on daily activities), 5 (Very severe problem, markedly influences daily activities or requires rest or both). The total minimum value is 4 and maximum value is 20. Higher score means worse outcome.
Adverse events | Through study completion, an average of 1 year
  Patient reported adverse events will be documented
Persistence of symptom improvement or recurrence of dyspeptic symptoms | At week 12 after randomization
  After 8 weeks of active intervention, all three groups will be kept on first line treatment only for additional 4 weeks. Persistence of symptom improvement or recurrence of four dyspeptic symptoms (Postprandial fullness, Early Satiety, Epigastric pain, Epigastric burning) after discontinuation of neuromodulators (amitriptyline and trifluoperazine) will be assessed and compared by a 5-point Likert Scale. The four main symptoms of dyspepsia, each will be graded as 1 (No problem), 2 (Mild problem, can be ignored when not thinking about it), 3 (Moderate problem, cannot be ignored but does not influence daily activities), 4 (Severe Problem, influences concentration on daily activities), 5 (Very severe problem, markedly influences daily activities or requires rest or both). The total minimum value is 4 and maximum value is 20. Higher score means worse outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Dhaka Medical College, Dhaka, Bangladesh